CLINICAL TRIAL: NCT06673160
Title: Pumping to Up Maternal Milk Production for Preterms (PUMMPP)
Brief Title: Pumping to Up Maternal Milk Production for Preterms
Acronym: PUMMPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Folasade Aderibigbe, Fellow Physician, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-300013718
Record Dates: First submitted 2024-10-23; First posted 2024-11-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breastfeeding; Breastmilk Expression
Keywords: breastmilk supply in preterm infant; breastfeeding preterm infants
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pumping every 2 hours (Experimental): Mothers of patients in this group will be assigned to pump/ express breastmilk every 2 hours.
  Interventions: Behavioral: Pumping every 2 hours
- Pumping every 3 hours (Active Comparator): Mothers of patients in this group will be assigned to pump/ express breastmilk every 3 hours.
  Interventions: Behavioral: breast pumping every 3 hours

INTERVENTIONS:
Behavioral: Pumping every 2 hours — The intervention will be pumping every 2 hours.
  Other Names: breast pumping every 2 hours
  Arms: Pumping every 2 hours
Behavioral: breast pumping every 3 hours — The intervention will be pumping every 3 hours
  Arms: Pumping every 3 hours

SUMMARY:
The goal of this clinical trial is to learn about the effect of breast-pumping frequency on breast milk supply/ volume in mothers of preterm infants. The main question it aims to answer is:

- What effect does pumping frequency have on breast milk supply.

Researchers will compare breastmilk supply of mothers who pump every 2 hours to the supply of those who pump every 3 hours to see if there is a difference in the amount of breastmilk they produce.

Participants will be assigned to either pump every 2 hours or every 3 hours and record how many milliliters of breastmilk they produce daily for the first 28 days of their baby's life.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants <32 weeks gestation
* Out-born infants transferred to our facility <48hours of life
* Infants <1500 grams at birth
* Infants whose parents/ guardians have provided legal consent for study participation

Exclusion Criteria:

* Infants with birthing persons' that are severe/critically ill
* Birthing persons of infants <18 years old
* Infants with terminal illness or decision to withhold or limit support
* infants with major congenital anomalies, chromosomal disorders, or congenital infections

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Volume of expressed breastmilk | From enrollment to 28 days of life
  The primary outcome measure will be the volume of expressed breastmilk obtained in mL per day in the group pumping every 2 hours compared the group pumping every 3 hours

SECONDARY OUTCOMES:
The percentage of donor breast milk feedings | From enrollment to 28 days of life
  This outcome will assess the percentage of any enteral feeding that is derived from donor breast milk.
The number of days alive on full feedings | From enrollment to 28 days of life
  The total number of days the infant received full enteral feeds (≥120 milliliters(mL)/kilogram(kg)/day).
The time to full feedings | From enrollment to 28 days of life
  The number of days it takes to initially reach full enteral feeds (≥120mL/kg/day)
The number of infants with clinical evidence of feeding intolerance | From enrollment to first 28 days after birth
  Infants that have enteral feeds withheld, or in other words made "nothing by mouth" (NPO) > 24 hours for feeding or abdominal issues
Number of central line days | In the first 28 days of life
  The total number of days the infant maintained any type of central line access.
The number of infants receiving any volume of breastmilk at time of discharge | From enrollment to hospital discharge
  Infants who are still receiving any volume of expressed breastmilk upon discharge will be identified and noted.
The number of infants exclusively feeding breastmilk at discharge | From enrollment to hospital discharge
  Whether or not enrolled infants are receiving all their nutrition from their mom's own expressed breastmilk upon discharge will be noted
Average change in weight | from birth to 36 weeks' corrected gestational age
  Changes in weight measured in grams (g) from birth to 36 weeks corrected gestational age
Average change in length | from birth to 36 weeks corrected gestational age
  Changes in length measured in centimeters (cm)
Average change in head circumference | from birth to 36 weeks' corrected gestational age
  Change in head circumference measured in centimeters (cm)
The Bayley Scales of Infant and Toddler Development (BSID) | from 18-26 months of age
  The Bayley's cognitive component composite score will be assessed and noted.
  The cognitive composite score is determined by comparing the child's performance to a normative age-matched sample defined by the assessment. They are interpreted as follows:
  Mean score of 100 (Standard deviation=15) at the 50th percentile signifies mid-average functioning.
  Scores below 85 (1 Standard deviation below the mean), at the 16th percentile, indicate mild impairment of being 'at risk' of developmental delay. Monitoring is recommended, along with advice to parents on techniques to enhance development or referral to a therapist based on the level of impairment.
  Score below 70 (2 Standard deviation below the mean), at the second percentile, indicate moderate to severe impairment.
  In general, scores falling in the lowest 10th percentile indicate developmental delay.
The Bayley Scales of Infant and Toddler Development (BSID) | From 18-26 months of age
  The Bayley's motor component composite score will be assessed and noted.
  The motor composite score is determined by comparing the child's performance to a normative age-matched sample defined by the assessment. They are interpreted as follows:
  Mean score of 100 (Standard deviation=15) at the 50th percentile signifies mid-average functioning.
  Scores below 85 (1 Standard deviation below the mean), at the 16th percentile, indicate mild impairment of being 'at risk' of developmental delay. Monitoring is recommended, along with advice to parents on techniques to enhance development or referral to a therapist based on the level of impairment.
  Score below 70 (2 Standard deviation below the mean), at the second percentile, indicate moderate to severe impairment.
  In general, scores falling in the lowest 10th percentile indicate developmental delay.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Travers CP, Carlo WA, McDonald SA, Das A, Ambalavanan N, Bell EF, Sanchez PJ, Stoll BJ, Wyckoff MH, Laptook AR, Van Meurs KP, Goldberg RN, D'Angio CT, Shankaran S, DeMauro SB, Walsh MC, Peralta-Carcelen M, Collins MV, Ball MB, Hale EC, Newman NS, Profit J, Gould JB, Lorch SA, Bann CM, Bidegain M, Higgins RD; Generic Database and Follow-up Subcommittees of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Racial/Ethnic Disparities Among Extremely Preterm Infants in the United States From 2002 to 2016. JAMA Netw Open. 2020 Jun 1;3(6):e206757. doi: 10.1001/jamanetworkopen.2020.6757. PMID 32520359
- [Background] Santoli CMA, Taylor-Cho IA, Darling AJ, Montoya MN, Gilner JB, Wheeler SM, Dotters-Katz SK. Predictors of Breastfeeding among Patients Admitted with Preterm Prelabor Rupture of Membranes. Am J Perinatol. 2024 May;41(S 01):e3196-e3201. doi: 10.1055/a-2211-1787. Epub 2023 Nov 15. PMID 37967869
- [Background] Quintero SM, Strassle PD, Londono Tobon A, Ponce S, Alhomsi A, Maldonado AI, Ko JS, Wilkerson MJ, Napoles AM. Race/ethnicity-specific associations between breastfeeding information source and breastfeeding rates among U.S. women. BMC Public Health. 2023 Mar 17;23(1):520. doi: 10.1186/s12889-023-15447-8. PMID 36932332
- [Background] Huang Y, Liu Y, Yu XY, Zeng TY. The rates and factors of perceived insufficient milk supply: A systematic review. Matern Child Nutr. 2022 Jan;18(1):e13255. doi: 10.1111/mcn.13255. Epub 2021 Aug 12. PMID 34382733
- [Background] Meek JY, Tippins S, American Academy of Pediatrics. American Academy of Pediatrics new mother's guide to breastfeeding. New York: Bantam Books; 2002. xiv, 258 p. p.